CLINICAL TRIAL: NCT01030354
Title: Effects of Protein-Enriched Meal on Liver, Kidney or Bone: a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Herbalife International of America, Inc. (Industry)
Responsible Party: Zhaoping Li, MD, PhD, Professor of Medicine, UCLA Center for Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCLA OPRS 03-06-120
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Weight Reduction; Obesity; Weight Management
Keywords: Satiety; Meal Replacements; High Protein; Standard Protein
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Intervention and Higher protein meal replacement (Active Comparator): A higher protein meal replacement diet based on 1 gram of protein per pound of lean body mass
  Interventions: Dietary Supplement: Herbalife Meal Replacements
- Dietary Intervention and Standard Protein Meal Replacement (Active Comparator): Standard protein meal replacement diet based on ½ gram of protein per pound of lean body mass
  Interventions: Dietary Supplement: Herbalife Meal Replacements

INTERVENTIONS:
Dietary Supplement: Herbalife Meal Replacements — Higher protein meal replacement diet based on 1 gram of protein per pound of lean body mass will improve weight loss in comparison to a standard protein meal replacement diet based on ½ gram of protein per pound of lean body mass
Dietary Supplement: Herbalife Meal Replacements — Higher protein meal replacement diet based on 1 gram of protein per pound of lean body mass will improve weight loss in comparison to a standard protein meal replacement diet based on ½ gram of protein per pound of lean body mass.

SUMMARY:
This study will examine whether a higher protein meal replacement diet (consisting of 1 gram of protein per pound lean body mass) is more effective in causing weight loss compared to a standard meal replacement protein diet (consisting of ½ gram of protein per pound of lean body mass). The study will assign approximately 100 subjects (50 each) to the following arms 1) higher meal replacement diet program 2) standard meal replacement diet program. All participants will meet with a registered dietitian to provide nutrition education and behavior modification, including general exercise recommendations. As part of your participation, you must be willing to undergo a measurement of body fat, and blood tests, and be willing to use Herbalife Meal replacements as part of your diet for the duration of the study (one year).

DETAILED DESCRIPTION:
There is concern that excess protein intake may be damaging to liver, renal function, and bone health. This study was designed to compare the effects of a high protein (HP) and an isocaloric meal standard protein (SP) weight loss plan on liver function, renal function and bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 years and older at screening
2. Female subjects must have a negative pregnancy test at screening, must be surgically sterile or at least 6 months postmenopausal or must use a form of birth control measure. Hormonal birth control, IUD, or abstinence will be acceptable as birth control measures. Other types of birth controls such as condom, diaphragm, or sponges may not be considered adequate forms of birth control measures in this study.
3. BMI of 27 to 40 kg/m2 inclusive.
4. Subjects must be in good health as determined by medical history, physical examination, and screening clinical laboratory including chemistry panel and CBC.

h. Must have stable smoking habits (or be non-smokers) for at least 6 months prior to screening and agree not to intend to change such habits during the course of the study.

i. Subjects requiring the regular use of any prescription medication may be admitted to the study providing the dose is stable.

j. Ethical

Subject must sign the Institutional Review Board-approved written informed consent prior to he initiation of any study specific procedures or randomization. A subject will be excluded for any condition that might compromise the ability to give truly informed consent for participation in the study.

Exclusion Criteria:

1. Weight Stability. Any subject who reports weight change of > 3.0 kg in the month prior to screening.
2. Any subject who has been on a very low calorie diet ( < 800 kcal/day) for a period of 4 months or more in the 12 months prior to screening, or who has lost > 10 kg in the 6 months prior to screening.
3. Use of any other investigational drug (s) within 8 weeks prior to screening.
4. Abnormal laboratory parameters: Serum creatinine > 1.6 mg/dl, Liver function tests, ALT, AST, Bili results > 2.0 times the upper limit of normal. Triglycerides > 500 mg/dl, total cholesterol > 350 mg/dl, TSH outside of normal range.
5. Subjects who drink more than 1 alcoholic beverages per day.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-07; Primary Completion 2005-07 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change in weight. | Baseline, 3, 6 and 12 months

SECONDARY OUTCOMES:
Secondary endpoints are changes in fasting plasma glucose levels associated with weight loss, insulin, blood pressure, lipid levels and body fat. | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Li Z, Treyzon L, Chen S, Yan E, Thames G, Carpenter CL. Protein-enriched meal replacements do not adversely affect liver, kidney or bone density: an outpatient randomized controlled trial. Nutr J. 2010 Dec 31;9:72. doi: 10.1186/1475-2891-9-72. PMID 21194471